CLINICAL TRIAL: NCT06619288
Title: Good-first: a Multicohort Study of B/F/TAF As First-line ART in a Public Hospital in Eastern China
Brief Title: Good-first: B/F/TAF As First-line ART
Status: Recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Nantong Third Peoples Hospital (Unknown)
Responsible Party: Principal Investigator, Gang Qin, MD, PhD, Associate Professor, Affiliated Hospital of Nantong University
Other Study IDs: 2024-TDF-058
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: HIV Infection
Keywords: B/F/TAF; TDF+3TC+EFV; DTG/3TC; Cohort study
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (6):
- HIV early presenters (TDF+3TC+EFV): 100 HIV-infected early presenters diagnosed between Jan 2020 and Jun 2023.
  Interventions: Drug: TDF+3TC+EFV
- HIV late presenters (TDF+3TC+EFV): 100 HIV-infected late presenters diagnosed between Jan 2020 and Jun 2023.
  Interventions: Drug: TDF+3TC+EFV
- HIV early presenters(DTG/3TC): 100 HIV-infected early presenters diagnosed between Jan 2020 and Jun 2023.
  Interventions: Drug: DTG/3TC
- HIV late presenters (DTG/3TC): 100 HIV-infected late presenters diagnosed between Jan 2020 and Jun 2023.
  Interventions: Drug: DTG/3TC
- HIV early presenters (B/F/TAF): 115 HIV-infected early presenters diagnosed between Jul 2024 and Jun 2025.
  Interventions: Drug: B/F/TAF
- HIV late presenters (B/F/TAF): 115 HIV-infected late presenters diagnosed between Jul 2024 and Jun 2025.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — Take one tablet per dose, once daily. Each tablet contains bictegravir (BIC) 50 mg, emtricitabine (FTC) 200 mg, and tenofovir alafenamide (TAF) 25 mg.
  Groups: HIV early presenters (B/F/TAF); HIV late presenters (B/F/TAF)
Drug: TDF+3TC+EFV — Take five tablets per dose, once daily. Each dose contains one tablet of tenofovir (TDF) 300 mg, one tablet of lamivudine (3TC) 300 mg, and three tablets of efavirenz (EFV) 200 mg (totaling 600 mg).
  Groups: HIV early presenters (TDF+3TC+EFV); HIV late presenters (TDF+3TC+EFV)
Drug: DTG/3TC — Take one tablet per dose, once daily. Each tablet contains dolutegravir (DTG) 50 mg and lamivudine (3TC) 300 mg.
  Groups: HIV early presenters(DTG/3TC); HIV late presenters (DTG/3TC)

SUMMARY:
This is a multicohort study conducted at Affiliated Hospital of Nantong University, and Nantong Third Peoples Hospital (Designated Hospital for HIV/AIDS Treatment of Nantong City), China. The study would involve 630 patients initiating HIV treatment, divided into six cohorts. The enrollment period for the prospective cohort is from July 2024 to June 2025, while the enrollment period for the retrospective cohort is from January 2020 to June 2023.

DETAILED DESCRIPTION:
Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) is recommended for initiating antiretroviral therapy (ART) in newly diagnosed HIV patients, including those with advanced disease. However, clinical data for this group is limited, and the high cost of B/F/TAF may hinder its widespread use as a first-line treatment.

This study aim to gather real-world evidence on the clinical practice of B/F/TAF as a first-line ART and address the knowledge gap regarding its cost-effectiveness. A multicohort study at the Designated Hospital for HIV/AIDS Treatment of Nantong City, China, involves 630 patients initiating HIV treatment, divided into six cohorts. There are 230 prospective patients on B/F/TAF (115 late presenters with CD4; 350 cells/μL or an AIDS-defining event, and 115 early presenters). Additionally, there are 400 retrospective patients on either tenofovir+lamivudine+efavirenz (TDF+3TC+EFV, 100 for each presentation group) or dolutegravir/lamivudine (DTG/3TC, 100 for each presentation group). The enrollment period for the prospective cohort is from July 2024 to June 2025, while the enrollment period for the retrospective cohort is from January 2020 to June 2023.

Data will be collected at baseline and at specific intervals over 48 weeks using electronic health records and patient-reported outcomes. Clinical data include time from diagnosis to ART initiation, plasma viral load (VL), CD4 count, adverse events, treatment adherence, and quality of life (QoL). QoL improvements will be assessed through questionnaires. Cost data will be collected following healthcare reporting standards. A microsimulation model will be adapted. The cost-effectiveness of B/F/TAF, compared to the other regimens, will be evaluated using clinical cohort data and modeling techniques to project long-term economic outcomes.

This study was approved by the ethics committee of Nantong Third Peoples Hospital. Consent will also be obtained from the participants during the study process.

This study followed the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) reporting guideline for cohort studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) diagnosed with HIV/AIDS, ART-naive, from July 2024 to June 2025 (prospective) or January 2020 to June 2023 (retrospective).
2. Eligible for ART initiation with B/F/TAF or previously treated with TDF+3TC+EFV or DTG/3TC.
3. Willing to adhere to study procedures and follow-up visits or have complete electronic health records (EHRs).

Exclusion Criteria:

1. Severe renal impairment (creatinine clearance < 50 mL/min).
2. Hepatitis B co-infection or severe hepatic impairment (Child-Pugh Class C).
3. Active tuberculosis (TB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of HIV-infected patients, including those who present in the early stages of infection as well as those with late-stage or advanced presentations. These individuals will encompass a wide range of clinical scenarios to ensure the findings are applicable to diverse patient populations.
Sampling Method: Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with virologic suppression | At 12 weeks, 24 weeks, and 48 weeks from the initiation of ART.
  Virologic suppression is defined as a plasma viral load (HIV RNA) of less than 50 copies/mL.
Change of CD4 count | At 12 weeks, 24 weeks, and 48 weeks from the initiation of ART.
  The percentage change in CD4+ T cell count from baseline after initiating ART, stratified by patients with lower versus higher baseline CD4+ levels.
Rate of immune reconstitution in late presenters | At 48 weeks from the initiation of ART.
  Immune reconstitution is defined as an immunological response in HIV late presenters, characterized by a CD4+ T cell count increase of at least 20% from baseline or reaching at least 350 cells/μL at 48 weeks, accompanied by an undetectable viral load.

SECONDARY OUTCOMES:
Rate of treatment discontinuation | From the initiation of ART until the end of the study, with an estimated period of assessment up to 104 weeks. This period includes monitoring from the date of ART initiation until the date of treatment discontinuation or study end.
  Throughout the entire follow-up period, there were instances of loss to follow-up or death due to other illnesses. If a subject experiences significant adverse reactions after taking the medication, it is necessary to discontinue the medication.
Number of adverse events | From the initiation of ART until the end of the study, with an estimated period of assessment up to 104 weeks. This period includes monitoring from the date of ART initiation until the date of treatment discontinuation or study end.
  Adverse events are mainly divided into five categories: central nervous system symptoms, which include headache, dizziness, insomnia, difficulty concentrating, mood changes, or mental confusion; gastrointestinal symptoms, such as nausea, vomiting, diarrhea, abdominal pain, or dyspepsia; hematologic symptoms, which involve low levels of red blood cells or hemoglobin, leading to fatigue, weakness, or pallor; hepatotoxicity, indicated by elevated liver enzyme levels, jaundice, or other signs of liver dysfunction; and dermatitis, which includes rash, itching, erythema, or dry skin.
QoL assessment | Assessed at baseline, and at 12, 24, and 48 weeks.
  Quality of Life (QoL) is assessed using the EQ-5D-5L scale, a standardized instrument developed by the EuroQol Group. It measures general health across five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with five levels of severity each. The index score ranges from -0.59 to 1, with higher scores indicating better health status.
HIV symptom assessment | Assessed at baseline, and at 12, 24, and 48 weeks.
  The HIV Symptom Index (HIV-SI) is used to assess the prevalence and severity of HIV-related symptoms. Scores range from 0 to 80, with higher scores indicating a greater burden of symptoms.
Mental health assessment | Assessed at baseline, and at 12, 24, and 48 weeks.
  People living with HIV (PLHIV) have a risk of experiencing depressive symptoms that is three times higher than that of the general population. The Patient Health Questionnaire-9 (PHQ-9), a self-administered scale, is used for diagnosing and monitoring depression. Scores on the PHQ-9 range from 0 to 27, with higher scores indicating more severe levels of depression. If a patient presents with moderate depressive symptoms (PHQ-9 score &gt; 9), he or she will be referred to a psychiatrist.
Cardiovascular risk assessment | Assessed at baseline, and at 12, 24, and 48 weeks.
  Cardiovascular risk assessment is an essential component of clinical practice for people living with HIV (PLHIV). The Framingham Risk Score is used to estimate the 10-year cardiovascular risk of an individual. Scores range from 0% to 30% or higher, with higher scores indicating a greater cardiovascular risk.

OTHER OUTCOMES:
Change of body weight | At 12 weeks, 24 weeks and 48 weeks from the initiation of ART.
  This metric represents the percentage change in body weight from the baseline measurement.
Change of LDL | At 12 weeks, 24 weeks and 48 weeks from the initiation of ART.
  Monitoring changes in low-density lipoprotein (LDL) cholesterol levels helps assess cardiovascular risk and the impact of ART on lipid profiles over time.
Change of eGFR | At 12 weeks, 24 weeks and 48 weeks from the initiation of ART.
  Estimated glomerular filtration rate (eGFR) calculated using serum creatinine levels is used to assess kidney function over time and indicates how well the kidneys are filtering waste from the blood. Changes in eGFR can signal improvements or declines in renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Qin, MD, PhD, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Nantong Third Peoples Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No